CLINICAL TRIAL: NCT01168076
Title: Noninvasive Transcutaneous Glucometer Development
Status: Completed | Type: Observational
Sponsor: InLight Solutions (Industry)
Responsible Party: Jeff Way, InLight Solutions
Other Study IDs: ILS-01-007
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2008-02

CONDITIONS: Healthy; Prediabetic State (IGT); Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The objective of this study is to assist in the development of a noninvasive device for the accurate measurement of blood glucose levels.

DETAILED DESCRIPTION:
The feasibility of measuring blood glucose concentration in patients with diabetes mellitus using near infrared (NIR) spectroscopy and multivariate data analysis techniques has been established using general purpose, scientific-grade infrared spectrophotometers under the 90-049 UNM HRRC protocol. Now that the concept of painless, bloodless, and reagent-less clinical laboratory tests has been shown to be viable, the challenge is to bring this technology to the patients who need it. We must develop a device that is portable, affordable, and rugged - all while improving accuracy. We must also improve our understanding of the nature of glucose in whole, intact skin. Since the light beam cannot discriminate plasma glucose in skin blood vessels from glucose in the larger skin interstitial fluid space, the exact nature of the glucose in all tissue compartments contributing to the light-beam signal must be elucidated. The noninvasive measurement can be no more accurate than the reference measurement on which it was based. Finally, we have found that the accuracy of the noninvasive measurement also worsens as a function of time from the initial measurement. This effect is independent of instrumentation drift and is due to physical changes in the patient's skin such as variation of hydration, collagen, vascularity, glycation end-products, etc. To account for these sources of physiologic interference they must be evaluated independently and then compared to errors of the noninvasive predictions over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Healthy
* Type I diabetics
* Type II diabetics
* Impaired glucose tolerance

Exclusion Criteria:

* Minor status (<18 years of age)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with Type 1 and 2 diabetes
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2001-12; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rohrscheib, M.D., Principal Investigator — UNMHSC
Locations (1):
- InLight Solutions, Albuquerque, New Mexico, United States

REFERENCES:
- See also: Related Info — http://www.inlightsolutions.com